CLINICAL TRIAL: NCT04444024
Title: Effect of Hypercholesterolemia Alone or Combined With Hypertension on the Degree of Coronary Artery Stenosis in Patients With Coronary Heart Disease Angina Pectoris: a Retrospective Study
Brief Title: Effect of Hypercholesterolemia With or Without Hypertension on Coronary Artery Stenosis in Patients With Angina: a Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunquan Yu, researcher, Tianjin University of Traditional Chinese Medicine
Other Study IDs: 2020TJUTCM
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Atherosclerotic Heart Disease With Angina Nos

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- NTC/-HTN group: Patients with TC < 5.18 mmol/l, systolic blood pressure <130 mmHg and diastolic blood pressure <80 mmHg belong to normal TC/ none hypertension(NTC/-HTN) group.
- NTC/+HTN group: Patients with TC < 5.18 mmol/l, systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥80 mmHg belong to normal TC/ hypertension(NTC/+HTN) group.
- BHTC/-HTN group: Patients whose TC is 5.18 ≤ TC < 6.19 mmol/l, systolic blood pressure <130 mmHg and diastolic blood pressure <80 mmHg belong to borderline-high TC/ none hypertension (BHTC/-HTN) group.
- BHTC/+HTN group: Patients whose TC is 5.18 ≤ TC < 6.19 mmol/l, systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥80 mmHg belong to borderline-high TC/ hypertension (BHTC/+HTN) group.
- HTC/-HTN group: Patients with TC ≥6.19 mmol/l, systolic blood pressure <130 mmHg and diastolic blood pressure <80 mmHg belong to high TC/ none hypertension(HTC/-HTN) group.
- HTC/+HTN group: Patients with TC ≥6.19 mmol/l, systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥ 80 mmHg belong to high TC/ hypertension(HTC/+HTN) group.

SUMMARY:
A multicenter, retrospective clinical study was carried out in the medical records management system of 6 hospitals in Tianjin. Patients who were suffered with Coronary heart disease angina pectoris and underwent coronary angiography are collected. The investigators collect and analyze the demographics, laboratory information, clinical outcome data, and coronary angiographic data of patients. To explore the correlation between hypercholesterolemia and the degree of coronary artery stenosis of Coronary heart disease angina pectoris, and to further research the influence of hypertension on total cholesterol level and coronary artery stenosis, and provide guidance for clinical prevention and treatment.

DETAILED DESCRIPTION:
Based on the total cholesterol level, the investigators divided patients into 3 groups: patients with TC < 5.18 mmol/l belong to normal TC (NTC) group, 5.18 ≤ TC < 6.19 mmol/l is borderline-high TC (BHTC) group, those with TC ≥6.19 mmol/l belong to high TC (HTC) group, and the correlation between the TC and the degree of coronary artery stenosis is evaluated. With or without hypertension will be further stratified to assess the effect of with or without hypertension on the correlation between TC levels and the degree of coronary artery stenosis. The 6 subgroups are: NTC/-HTN group, NTC/+HTN group, BHTC/-HTN group, BHTC/+HTN group, HTC/-HTN group, HTC/+HTN group.

The investigators refer to the recent diagnostic guidelines for coronary heart disease angina pectoris at home and abroad. The diagnosis can be given if it meets any one or more of the following:

1. There was a clear history of old myocardial infarction.
2. Previous coronary angiography or coronary CTA examination showed that at least one major branch of coronary artery has a lumen diameter stenosis ≥50%.
3. Those with ST-segment depression or T-wave inversion on ECG after coronary revascularization.

The investigators will redefined hypertension as systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥80 mmHg according to the recently published 2017 ACC/AHA guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 35 to 75 years old, male or female.
2. Those who were hospitalized between September 1, 2014 and September 1, 2019.
3. Patients with Coronary heart disease angina pectoris and have undergone coronary angiography in the inpatient department of cardiovascular internal medicine.
4. The diagnosis of hypercholesterolemia, Coronary heart disease angina pectoris and hypertension is accorded with the diagnostic criteria.

Exclusion Criteria:

1. Those with other cardiac diseases, gastroesophageal reflux disease or hiatal hernia, neurosis, spinal or vertebral artery cervical spondylosis, hyperthyroidism, climacteric syndrome, etc.
2. Those with myocarditis, cardiomyopathy, acute myocardial infarction, third degree of heart failure, severe heart valve disease, major diseases such as malignant tumor and serious metabolic diseases, liver failure or renal failure.
3. Those with psychotic disorders, or cognitive dysfunction.
4. Those of childbearing age and have fertility requirements, or pregnant women or lactating women.
5. Those allergic to iodine contrast medium.
6. Those who are not suitable for the study, as judged by the researcher.

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The collaborative network of Coronary heart disease research medical units formed by the research team includes the First affiliated Hospital of Tianjin University of traditional Chinese Medicine, the Second affiliated Hospital of Tianjin University of traditional Chinese Medicine, Tianjin Nankai Hospital, the affiliated Hospital of Tianjin Institute of traditional Chinese Medicine, Tianjin chest Hospital and Tianjin Medical University General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose in clinical biochemical tests. | one year
  In the hospital medical record management system, the investigators collect the fasting blood glucose data of the first day of hospitalization of the patients.
Glycated hemoglobin in clinical biochemical tests. | one year
  In the hospital medical record management system, the investigators collect the glycated hemoglobin data of the first day of hospitalization of the patients.
Total cholesterol in clinical biochemical tests. | one year
  In the hospital medical record management system, the investigators collect the total cholesterol data of the first day of hospitalization of the patients.
Triglyceride in clinical biochemical tests. | one year
  In the hospital medical record management system, the investigators collect the triglyceride data of the first day of hospitalization of the patients.
Low density lipoprotein cholesterol in clinical biochemical tests. | one year
  In the hospital medical record management system, the investigators collect the low density lipoprotein cholesterol data of the first day of hospitalization of the patients.
High density lipoprotein cholesterol in clinical biochemical tests. | one year
  In the hospital medical record management system, the investigators collect the high density lipoprotein cholesterol data of the first day of hospitalization of the patients.
C-reactive protein in clinical biochemical tests. | one year
  In the hospital medical record management system, the investigators collect the C-reactive protein data of the first day of hospitalization of the patients.
Fibrinogen in clinical biochemical tests. | one year
  In the hospital medical record management system, the investigators collect the fibrinogen data of the first day of hospitalization of the patients.
Coronary angiography data in imaging examination. | one year
  In the hospital medical record management system, the investigators collect coronary angiography data of the patient's hospitalization.
Age in demographics. | one year
  In the hospital medical record management system, the investigators collect the age data of the first day of hospitalization of the patients.
Gender in demographics. | one year
  In the hospital medical record management system, the investigators collect the gender data of the first day of hospitalization of the patients.
Ethnicity in demographics. | one year
  In the hospital medical record management system, the investigators collect the ethnicity data of the first day of hospitalization of the patients.
Weight in demographics. | one year
  In the hospital medical record management system, the investigators collect the weight data of the first day of hospitalization of the patients.
Smoking in demographics. | one year
  In the hospital medical record management system, the investigators collect the smoking data of the first day of hospitalization of the patients.
Medical history in demographics. | one year
  In the hospital medical record management system, the investigators collect the medical history data of the first day of hospitalization of the patients.
Blood pressure in demographics. | one year
  In the hospital medical record management system, the investigators collect the blood pressure data of the first day of hospitalization of the patients.

SECONDARY OUTCOMES:
Evaluate the correlation between total cholesterol level and the degree of coronary artery stenosis | one year
  Based on the total cholesterol level, the investigators divide patients into 3 groups. According to the location and degree of the lumen stenosis, the score of the degree of each coronary artery stenosis is calculated.
Assess the effect of with or without hypertension on the correlation between total cholesterol level and the degree of coronary artery stenosis | one year
  According to with or without hypertension, the patients are further divided into 6 subgroups.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes